CLINICAL TRIAL: NCT01155843
Title: Neural Mechanisms by Which Chronic Stress Regulates Inflammation in Asthma
Brief Title: Neural Mechanisms in Asthma
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: K01AT006202 (NIH)
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2014-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asthmatic, chronic stress
- Asthmatic, non-stress

SUMMARY:
Asthma is a chronic disease that affects nearly 13% of adults in the U.S., causing substantial impairment that is reflected in the tens of millions of missed days of work, and doctors' and emergency room visits it leads to annually. Those who have asthma are twice as likely to develop depression and anxiety, which are associated with more frequent and severe asthma symptoms, especially in those under chronic stress. The project proposed here seeks to understand the role of the brain in these associations and to evaluate the neural mechanisms through which a safe, low-cost intervention, that influences the function of body via the mind, may diminish the expression of asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatics:

  * Physician diagnosed asthma with previous use of asthma medication
* Controls:

  * negative skin-prick test to cat dander or house dust mite and have no history of asthma
* Chronic Stress:

  * score 3 or above on any subscale of the UCLA (University of California Los Angeles) chronic stress interview

No chronic stress:

score 1.5 or below on all subscales of the UCLA chronic stress interview

Exclusion Criteria:

* Individuals with severe asthma, or those whom currently require the use of corticosteroids
* Individuals with significant medical problems
* Individuals who smoke cigarettes
* Individuals a previous adverse reaction to corticosteroids, a recent (< 1 month) viral illness, a history of severe asthma or anaphylaxis.
* Breastfeeding women or women who are, suspect they might be or are trying to become pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Neural activity in response to stress | duration of stress (30 minutes)
  positron emission tomography
inflammation | 24 hours
  infiltration of eosinophils into lung sputum, percentage of blood eosinophils, exhaled nitric oxide, glucocorticoid sensitivity of peripheral blood leukocytes
lung function | 24 hours
  peak expiratory volume in 1 sec effort
peripheral acute stress reactivity | 60 minutes
  salivary cortisol and alpha amylase in response to acute stressor

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States